CLINICAL TRIAL: NCT05754320
Title: Tension Band Wire Fixation Versus Plating for Simple Displaced Olecranon Fractures: A Long-Term Prospective Randomized Trial
Brief Title: TBW vs Plating in Olecranon Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Yonnatan Persitz, Principal Investigator, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 94/13
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Olecranon Fracture
MeSH Terms: conditions — Olecranon Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tension Band Wire fixation (Experimental): patients suffering simple olecranon fracture, randomized for treatment of tension band wire fixation
  Interventions: Device: Tension band wire fixation
- Plate fixation (Experimental): patients suffering simple olecranon fracture, randomized for treatment of plate fixation
  Interventions: Device: Plate fixation

INTERVENTIONS:
Device: Tension band wire fixation — Tension band wire fixation
  Arms: Tension Band Wire fixation
Device: Plate fixation — Tension band wire fixation
  Arms: Plate fixation

SUMMARY:
Background: While the tension band wiring (TBW) technique is commonly used for simple, displaced olecranon fractures, it is associated with complications such as hardware prominence. To date, studies comparing between the efficacy and safety of TBW and plate fixation for these fractures have not provided a conclusive answer.

Purposes: To investigate which of the two techniques provide better functional and radiological outcomes for simple displaced Mayo type 2A olecranon fractures, Which technique provides better patient-reported outcomes, What are the complication rates associated with each technique

DETAILED DESCRIPTION:
Background: While the tension band wiring (TBW) technique is commonly used for simple, displaced olecranon fractures, it is associated with complications such as hardware prominence. To date, studies comparing between the efficacy and safety of TBW and plate fixation for these fractures have not provided a conclusive answer.

Purposes: To investigate which of the two techniques provide better functional and radiological outcomes for simple displaced Mayo type 2A olecranon fractures, Which technique provides better patient-reported outcomes, What are the complication rates associated with each technique Methods: A long-term, prospective, randomized study on 50 adult patients who underwent surgery to treat acute, simple, displaced olecranon fractures in a Hand and Upper Extremity Surgery Unit at a tertiary care center between November 2012 and October 2017. Patients were randomized on a 1:1 basis to either tension band or plate fixation and were evaluated at 2 weeks, 6 weeks, 3 months, 6 months, and 1 year after surgery. Evaluation of long-term complications continued after 1 year as clinically indicated. The primary outcome measure was the 1-year postoperative Disabilities of the Arm, Shoulder and Hand (DASH) score. Additional outcome measures included patient-reported Oxford elbow score, functional (i.e., range of motion) and radiographic assessments and complication rates.

ELIGIBILITY:
Inclusion Criteria:

1. traumatic non-pathological simple olecranon fracture
2. age 18 years or older
3. presentation within 2 weeks of injury.

Exclusion Criteria:

1. inability to sign an informed consent
2. inability to comply with follow-up
3. associated elbow fractures
4. open fractures
5. pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11-10 (Actual); Primary Completion 2017-10-28 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand score | 1 year
  1-year postoperative patient reported Disabilities of the Arm, Shoulder and Hand score. Scale - 0 (no disability) to 100 (most severe disability)

SECONDARY OUTCOMES:
Oxford elbow score | 1 year
  1-year postoperative patient-reported Oxford elbow score. Scale - 0 (worst elbow functional score) to 48 (normal elbow functional score)
Union rate | 1 year
  Union rate
Complication rate | >1 year
  Long term complication rate

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Medical Center (Yitzhak Shamir Medical Center), Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No